CLINICAL TRIAL: NCT07295418
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Clinical Study to Evaluate the Safety and Efficacy of SAL003 Monotherapy in Participants With Hypercholesterolemia and Mixed Dyslipidemia
Brief Title: A Study of SAL003 in Participants With Hypercholesterolemia and Mixed Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Salubris (Chengdu) Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL003A301
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hyperlipidemias
Keywords: Low-density lipoprotein cholesterol; PCSK9; SAL003
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Drug: SAL003 140 mg
  Interventions: Drug: SAL003 140 mg
- Reference Group (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAL003 140 mg — Double-blind treatment period: Administer SAL003 140mg subcutaneously once every 4 weeks for a total of 3 times. Collect efficacy and safety results after 12 weeks. Extended administration period: Administer SAL003 140mg subcutaneously once every 4 weeks and follow up until 52 weeks to collect efficacy and safety results.
  Arms: Test Group
Drug: Placebo — Double-blind treatment period: Administer Placebo subcutaneously once every 4 weeks for a total of 3 times. Collect efficacy and safety results after 12 weeks. Extended administration period: Administer SAL003 140mg subcutaneously once every 4 weeks and follow up until 52 weeks to collect efficacy and safety results.
  Arms: Reference Group

SUMMARY:
This is a Phase 3 study to evaluate the efficacy and safety of SAL003, a fully human monoclonal antibody against PCSK9, as monotherapy in Chinese participants with hypercholesterolemia and mixed dyslipidemia. Participants who are not on lipid-lowering therapy or have washed out from previous therapy will be randomized in a 2:1 ratio to receive either SAL003 140 mg or matching placebo, administered subcutaneously every 4 weeks for 12 weeks. Following the double-blind period, all participants will enter an open-label extension period and receive SAL003 140 mg Q4W for an additional 40 weeks. The primary objective is to demonstrate the superiority of SAL003 over placebo in reducing Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, Phase 3 clinical trial. The study consists of four periods: a Screening Period (up to 1 week), a Run-in Period (2 weeks), a Double-blind Treatment Period (12 weeks), and an Extended Treatment Period (40 weeks), with a total study duration of approximately 55 weeks per participant.

Approximately 600 participants will be randomized. Eligible participants must be aged 18-75 years with a fasting LDL-C level between 2.6 mmol/L and 4.9 mmol/L, who are either statin-naïve or have washed out from lipid-lowering drugs for at least 3 months. Key exclusion criteria include familial hypercholesterolemia, established atherosclerotic cardiovascular disease (ASCVD), uncontrolled hypertension, poorly controlled diabetes, and significant hepatic or renal impairment.

In the Double-blind Period, participants will be stratified by baseline LDL-C (<3.4 mmol/L or ≥3.4 mmol/L) and randomized to receive either SAL003 140 mg or placebo via subcutaneous injection every 4 weeks for 3 doses (Days 1, 29, and 57). After completing the 12-week double-blind period, all participants will enter the Extended Treatment Period and receive open-label SAL003 140 mg Q4W for 10 additional doses (from Week 12 to Week 52).

The primary efficacy endpoint is the percent change from baseline in LDL-C at Week 12. Key secondary endpoints include the change from baseline in LDL-C at Week 12, the proportion of participants achieving LDL-C target goals at Week 12 and Week 52, and the percent change from baseline in other lipid parameters (e.g., TC, TG, Non-HDL-C, ApoB) at Week 12 and Week 52. Safety, immunogenicity, and pharmacokinetics will be assessed throughout the study.

The primary analysis will be performed on the Full Analysis Set (FAS) using a repeated measures mixed-effects model (MMRM) to compare the least-squares mean difference between the SAL003 and placebo groups at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 75 years (inclusive).
* Fasting LDL-C ≥2.6 mmol/L and <4.9 mmol/L at screening/randomization.
* Meets criteria based on the 2023 Chinese Lipid Management Guidelines (e.g., specific LDL-C levels with certain risk factors, or presence of diabetes).
* Fasting triglycerides (TG) ≤5.6 mmol/L at screening/randomization.
* Provides written informed consent.

Exclusion Criteria:

* Diagnosis of familial hypercholesterolemia (HoFH or HeFH).
* History of atherosclerotic cardiovascular disease (ASCVD).
* Uncontrolled hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg).
* Type 1 diabetes or poorly controlled Type 2 diabetes (HbA1c >8.0%).
* Significant hepatic or renal impairment.
* Active liver disease or positive for HIV or Syphilis.
* History of malignancy within 5 years prior to screening.
* Use of any lipid-lowering drugs (statins, ezetimibe, etc.) or traditional Chinese medicines known to affect lipid metabolism within 3 months prior to screening.
* Prior treatment with any PCSK9 inhibitor.
* Known hypersensitivity to any component of the investigational product or history of severe allergy to antibody therapies.
* Any other condition deemed by the investigator to be unsuitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Percent change of Low-Density Lipoprotein Cholesterol (LDL-C). | at Week 12
  Percent change from baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No